CLINICAL TRIAL: NCT01433146
Title: Effect of Temperament, Anxiety and Depression on Immuninity in Colorectal Cancer Patients.
Brief Title: Effect of Temperament, Anxiety and Depression on Immuninity in Colorectal Cancer Patients. Effetti Del Temperamento, Dell'Ansia e Della Depressione Sulla Sopravvivenza Globale e Sulla Risposta Immunitaria Del Paziente Affetto da Adenocarcinoma Colo-Rettale.
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Marco La Torre, Medical Doctor, PhD, University of Roma La Sapienza
Other Study IDs: 65422-SU-CE
Record Dates: First submitted 2011-09-10; First posted 2011-09-13 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Temperament; Anxiety; Depression; Colorectal Cancer
Keywords: Temperament; Anxiety; Depression; Colorectal Cancer
MeSH Terms: conditions — Anxiety Disorders; Depression; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for cell-mediated immunity evaluaion
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Aim of the study is to evaluate if Temperament, Anxiety and Depression can affect Immunity and influence Survival in Colorectal Cancer Patients

DETAILED DESCRIPTION:
120 prospective patients, with non-metastatic colorectal cancer, will be evaluated with questionnaires and auto-questionnaires in order to assess temperament, anxiety and depression. The immunity status will be assessed by a blood sample with the aim to evaluate cell-mediated immunity.

Survivall will be related to level of anxiety/temperament/depression and cell-mediated immunity.

Univariate and multivariate model analisys will be performed in order to evaluate if anxiety/temperament/depression and cell-mediated immunity can be considered as prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

diagnosis of non-metastatic colorectal cancer

Exclusion Criteria:

previous other primary malignancies immunodepression diagnosis of major deppression diagnosis of anxiety/depression syndrome

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Temperament in non-metastatic colorectal cancer patients | 24 months
  Evaluation if Temperament can be considered as dependent or indipendent prognostic factor for survival in non-metastatic colorectal cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Marco La Torre, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- "Sapienza" University of Rome, Rome, Rome, Italy

REFERENCES:
- [Background] Nan KJ, Wei YC, Zhou FL, Li CL, Sui CG, Hui LY, Gao CG. Effects of depression on parameters of cell-mediated immunity in patients with digestive tract cancers. World J Gastroenterol. 2004 Jan 15;10(2):268-72. doi: 10.3748/wjg.v10.i2.268. PMID 14716837
- [Background] Kohno Y, Maruyama M, Matsuoka Y, Matsushita T, Koeda M, Matsushima E. Relationship of psychological characteristics and self-efficacy in gastrointestinal cancer survivors. Psychooncology. 2010 Jan;19(1):71-6. doi: 10.1002/pon.1531. PMID 19204934